CLINICAL TRIAL: NCT03180294
Title: Phase II Double Blind Dose Finding Trial of Bupropion Versus Placebo for Sexual Desire in Women With Breast or Gynecologic Cancer
Brief Title: Bupropion Hydrochloride in Improving Sexual Desire in Women With Breast or Gynecologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NRG-CC004; NCI-2017-00344 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC004 (Other: NRG Oncology); NRG-CC004 (Other: DCP); UG1CA189867 (NIH)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Breast Carcinoma; Cervical Carcinoma; Ovarian Carcinoma; Postmenopausal; Uterine Corpus Cancer; Vaginal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bupropion 150 mg (Experimental): One Bupropion 150 mg XL capsule by mouth (PO) in a.m. daily for one week; one Bupropion 150 mg XL capsule and one placebo capsule daily for 8 weeks; one placebo capsule daily for one 1 week (titration off).
  Interventions: Drug: Bupropion 150 mg XL; Drug: Placebo
- Bupropion 300 mg (Experimental): One Bupropion 150 mg XL capsule PO in a.m. daily for one week; two Bupropion 150 mg XL capsules PO in a.m. daily for 8 weeks (300 mg target dose); one Bupropion 150 mg XL capsule PO in a.m. daily for 1 week (titration off)
  Interventions: Drug: Bupropion 150 mg XL
- Placebo (Placebo Comparator): One placebo capsule PO in a.m. daily for 1 week; two placebo capsules PO in a.m. daily for 8 weeks; one placebo capsule PO in a.m. daily for 1 week (titration off)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion 150 mg XL — By mouth
  Other Names: Amfebutamone; BUPROPION HYDROCHLORIDE; BW 323U66; Forfivo XL; Wellbutrin; Zyban
  Arms: Bupropion 150 mg; Bupropion 300 mg
Drug: Placebo — By mouth
  Arms: Bupropion 150 mg; Placebo

SUMMARY:
This phase II randomized trial studies how well bupropion hydrochloride works in improving sexual desire in women with breast or gynecological cancer. Bupropion hydrochloride may work by boosting sexual desire, energy, or motivation without causing intolerable or undesirable side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure the ability of two dose levels of bupropion hydrochloride (bupropion), 150 or 300 mg of extended release, to improve sexual desire more than a placebo at 9 weeks (8 weeks on the target dose) as measured by the desire subscale of the female sexual function index (FSFI).

SECONDARY OBJECTIVES:

I. Evaluate the side effects of 150 and 300 mg bupropion extended release and differentiate these side effects from those observed in the placebo arm.

II. Evaluate the effect of 150 and 300 mg of bupropion extended release on the Patient Reported Outcomes Measurement Information System (PROMIS) fatigue scale, PROMIS sexual desire and satisfaction measure, patient health questionnaire (PHQ)-4, and the FSFI total score, at 5 and 9 weeks, as well as the desire subscale score of the FSFI at 5 weeks.

III. Evaluate the effect of 150 and 300 mg of bupropion extended release on the global impression of change scale and the patient's perception of risk versus (vs.) benefit at 5 weeks (4 weeks at target dose) and 9 weeks (8 weeks at target dose).

Patients are randomized to 1 of 3 arms.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* Score of < 9 on the PHQ-4
* Patients must have a FSFI desire subscale baseline score less than 3.3

  * NOTE-Both the PHQ-4 and FSFI must be completed by the patient and data entered in Oncology Patient Enrollment Network (OPEN) at Step 1 registration to determine eligibility
* Diagnosis of breast or gynecologic cancer [examples are lobular carcinoma in situ (LCIS),ductal carcinoma in situ (DCIS), invasive breast, ovarian, endometrial, vulvar, cervical and vaginal]
* Completed definitive therapy consisting of surgery, chemotherapy or radiation therapy at least 180 days ago (may continue on Herceptin or endocrine therapy)
* Post menopausal as defined by at least ONE of the following:

  * 12 months (365 days) without a period;
  * Bilateral oophorectomy;
  * Chemically induced menopause as long as there are no plans to stop during the study;
  * For women 57 and under, if at least one ovary and woman has had hysterectomy, must have follicle stimulating hormone (FSH) (> 30 mIU/mL) and estradiol in menopausal range per institution?s laboratory (< 10 for ultra sensitive assay: < 25-30 otherwise);
  * At least one ovary intact and 180 days without a period with FSH (> 30 mIU/mL) and estradiol in menopausal range per institution's laboratory (< 10 for ultra sensitive assay: < 25-30 otherwise); Note: Women 58 and older do not have to have hormonal tests.
* History, physical and performance status of 2 or less within 180 days prior to registration
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Glomerular filtration rate > 90ml/min
* For breast cancer patients only, endocrine therapies are allowed (such as aromatase inhibitors, but not current tamoxifen. Prior tamoxifen is permitted with a 30 day wash out period). )
* Vaginal estrogen is allowed, for all protocol disease sites, if dose equal to or less than that in estring (< 7.5 mcg) and it has been used for at least 30 days with no plans to stop or alter use during the course of the study
* Antidepressants for mood and hot flashes, including selective serotonin reuptake inhibitors (SSRIs) will be allowed if patients have been on a stable dose for the last 60 days and the dose is not expected to change during the course of the study; only subthreshold or low dose antidepressants will be allowed (e.g. Effexor up to 75 mg or Lexapro 5-10 mg or Celexa 10- 20 mg)
* The patient must provide study-specific informed consent prior to study entry/screening
* Women who report that their motivation/desire for sexual intimacy has decreased since her cancer diagnosis
* Able to swallow whole capsules
* Proficient in English (due to number of questionnaires not validated in other languages)
* Completion of the FSFI and PHQ-4; both questionnaires will be required and data entered at the time of step 1 registration
* PRIOR TO STEP 2 RANDOMIZATION
* Completion of the following baseline quality of life forms: PHQ-4, FSFI, PROMIS sexual function and satisfaction, PROMIS fatigue short form 8a, Impact of Treatment Scale, patient reported outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) items, and revised dyadic adjustment scale; these quality of life forms will be required and data must be entered in Medidata Rave at step 2 registration; if available at the time of step 1 registration, step 2 registration can take place immediately after step 1; women who do not currently have a partner do not have to complete the revised dyadic adjustment scale; enter "no partner" for this form

Exclusion Criteria:

* Untreated depression, major depressive disorder (MDD), suicidal ideations or anxiety disorders in the past 5 years per the medical chart based on Diagnostic and Statistical Manual (DSM) IV diagnoses
* Seizure disorders
* Current or history of anorexia or bulimia in the past 5 years
* Allergy to bupropion
* Use of drugs metabolized by CYP2D6
* Stage IV cancer
* History of Parkinson's disease, multiple sclerosis or fibromyalgia
* Extensive pelvic exenteration surgery, surgeries which include partial or total vaginectomy with or without reconstruction; radical vulvectomy with or without remove of clitoris
* Women who are currently undergoing or planning to undergo reconstruction surgery during the course of the study; women who have completed reconstruction surgery must be 30 days from surgery
* Oral or transdermal estrogen therapy is not allowed
* Males are not permitted to participate
* Patients undergoing abrupt discontinuation of alcohol, benzodiazepines, barbiturates, and antiepileptic drugs after chronic use
* Patients who discontinue monoamine oxidase (MAO)-inhibitor (I)'s within 14 days prior to starting the investigational drug
* Poorly controlled hypertension (systolic blood pressure [BP] >= 160 mmHg or diastolic BP >= 100 mmHg) on three or more readings in the past 12 months
* Patients with active bipolar disorder
* Patients with impaired decision making as determined by the treating physician
* Concurrent use of bupropion
* Concomitant invasive malignancy requiring treatment other than non-melanomatous skin cancer.
* Previous or concurrent use of flibanserin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, Principal Investigator — NRG Oncology
Locations (362):
- United States (362):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Willis-Knighton Medical and Cancer Center, Shreveport, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Lenox Hill Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

REFERENCES:
- [Derived] Barton DL, Pugh SL, Ganz PA, Plaxe SC, Koontz BF, Carter J, Greyz-Yusupov N, Page SJ, Rowland KM Jr, Balcueva EP, Nabeel S, Basil JB, Hill ML, Muller CY, Bell MC, Deshmukh S, Kachnic LA. Randomized Controlled Phase II Evaluation of Two Dose Levels of Bupropion Versus Placebo for Sexual Desire in Female Cancer Survivors: NRG-CC004. J Clin Oncol. 2022 Feb 1;40(4):324-334. doi: 10.1200/JCO.21.01473. Epub 2021 Dec 9. PMID 34882500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Registered patients who completed required baseline assessments were randomized. Of 238 registered patients, 230 were randomized.
Groups:
- Bupropion 150 mg: One Bupropion 150 mg XL capsule by mouth (PO) in a.m. daily for one week; one Bupropion 150 mg XL capsule and one placebo capsule PO in a.m. daily for 8 weeks; one placebo capsule daily PO in a.m. for one 1 week (titration off).
Period: Overall Study
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Started | 79 | 74 | 77
Eligible Population | 79 | 74 | 77
Adverse Event Population (Eligible participants with adverse event data who started study treatment.) | 77 | 73 | 76
Completed (Participants contributing data to results are considered to have completed the study.) | 79 | 74 | 77
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Bupropion 300 mg: One Bupropion 150 mg XL capsule PO in a.m. daily for one week; two Bupropion 150 mg XL capsules PO in a.m. daily for 8 weeks (300 mg target dose); one Bupropion 150 mg XL PO in a.m. daily for 1 week (titration off)
- Total: Total of all reporting groups
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo | Total
Number analyzed (Participants) | 79 | 74 | 77 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.63 (7.61) | 54.68 (9.05) | 58.1 (8.00) | 55.8 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 74 | 77 | 230
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 11
  Not Hispanic or Latino | 74 | 69 | 72 | 215
  Unknown or Not Reported | 2 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 3 | 3 | 6
  White | 74 | 70 | 67 | 211
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 3 | 5
Zubrod [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death.
  Participants
    0 | 70 | 70 | 66 | 206
    1 | 9 | 4 | 11 | 24
Current Selective Serotonin Reuptake Inhibitors (SSRI) Use [Count of Participants; unit: Participants]
  No | 69 | 69 | 66 | 204
  Yes | 10 | 5 | 11 | 26
Prior Pelvic Radiation Therapy [Count of Participants; unit: Participants]
  No | 70 | 72 | 68 | 210
  Yes | 9 | 2 | 9 | 20
Prior Pelvic Surgery [Count of Participants; unit: Participants]
  No | 56 | 54 | 48 | 158
  Yes | 23 | 20 | 29 | 72
Aromatase Inhibitor therapy [Count of Participants; unit: Participants]
  No | 44 | 37 | 42 | 123
  Yes | 35 | 37 | 35 | 107

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 9 Weeks in the Desire Subscore of the Female Sexual Function Index ("Sexual Desire")
Description: The desire subscore of the female sexual function index (FSFI) measures self-reported sexual desire. Possible scores range from 1.2 to 6, with higher scores indicating increased desire. Change score is calculated by subtracting baseline from later score, with a positive change score indicating increased desire. This measure is referred to as "sexual desire" in the protocol.
Time Frame: Baseline (prior to randomization) and 9 weeks from start of study treatment (within 21 days of randomization)
Population: Eligible participants with baseline and 9 week data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 66 | 59 | 63
units on a scale | 0.64 (0.95) | 0.60 (0.89) | 0.62 (1.18)
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Using a two sample t-test with a one-sided type I error of 0.05 (overall type I error of 0.1 after a Bonferroni correction) and an effect size of 0.45, 62 patients/arm were calculated to be needed to achieve 80% statistical power. Adjusting for 20% non-compliance resulted in a total sample size of 234 patients; Test type: Superiority; p = 0.46, t-test, 1 sided
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.54, t-test, 1 sided

2. Secondary Outcome: Change From Baseline in the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Score
Description: The PROMIS fatigue score measures self-reported fatigue symptoms over the past 7 days. Possible scores range from 33.1 to 77.8, with higher scores indicating more fatigue. Change score is calculated by subtracting baseline from later score, with a positive change score indicating increased fatigue.
Time Frame: Baseline (prior to randomization) and 5 and 9 weeks from start of study treatment (within 21 days of randomization)
Population: Eligible with baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bupropion 150 mg: One Bupropion 150 mg XL capsule PO in a.m. daily for one week; one Bupropion 150 mg XL capsule and one placebo capsule PO in a.m. daily for 8 weeks; one placebo capsule daily PO in a.m. for one 1 week (titration off).
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 79 | 74 | 77
units on a scale
  Week 5: number analyzed (Participants) | 64 | 60 | 62
  Week 5 | -2.29 (7.05) | -1.11 (7.63) | -0.30 (6.71)
  Week 9: number analyzed (Participants) | 65 | 59 | 62
  Week 9 | -3.28 (9.46) | -3.14 (7.88) | -3.42 (6.59)
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Week 5; Test type: Superiority; p = 0.95, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; Week 5; Test type: Superiority; p = 0.73, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 3: Comparison: Bupropion 150 mg vs Bupropion 300 mg; Week 9; Test type: Superiority; p = 0.46, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 4: Comparison: Bupropion 150 mg vs Placebo; Week 9; Test type: Superiority; p = 0.42, t-test, 1 sided — One-sided significance level 0.05

3. Secondary Outcome: Change From Baseline at 5 Weeks in Desire Subscore of the FSFI ("Sexual Desire")
Description: as for outcome 1
Time Frame: Baseline (prior to randomization) and 5 weeks from start of study treatment (within 21 days of randomization)
Population: Eligible with baseline and 5 week data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 66 | 61 | 63
units on a scale | 0.70 (0.90) | 0.48 (0.69) | 0.58 (0.99)
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Test type: Superiority; p = 0.24, t-test, 1 sided — One-side significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 150 mg vs Placebo; Test type: Superiority; p = 0.74, t-test, 1 sided — One-sided significance level 0.05

4. Secondary Outcome: Change From Baseline in the PROMIS Global Satisfaction With Sex Life Subscore of Sexual Function and Satisfaction Measure ("Sexual Desire and Satisfaction")
Description: The PROMIS Global Satisfaction with Sex Life subscore measures self-reported global satisfaction, interest, and interference in sexual health over the past 7 days. Possible scores range from 3 to 30, with higher scores indicating more satisfaction with sex life. Change score is calculated by subtracting baseline from later score, with a positive change score indicating increased satisfaction. This score is referred to as the "PROMIS sexual desire and satisfaction measure" in the protocol.
Time Frame: Baseline (prior to randomization) and 5 and 9 weeks from start of study treatment (within 21 days of randomization)
Population: Eligible with baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 79 | 74 | 76
units on a scale
  Week 5: number analyzed (Participants) | 65 | 59 | 61
  Week 5 | 3.35 (7.27) | 2.81 (5.82) | 3.08 (6.00)
  Week 9: number analyzed (Participants) | 65 | 60 | 60
  Week 9 | 2.05 (6.51) | 2.72 (4.72) | 3.58 (6.93)
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Week 5; Test type: Superiority; p = 0.41, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; Week 5; Test type: Superiority; p = 0.60, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 3: Comparison: Bupropion 150 mg vs Placebo; Week 9; Test type: Superiority; p = 0.90, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 4: Comparison: Bupropion 300 mg vs Placebo; Week 9; Test type: Superiority; p = 0.79, t-test, 1 sided — One-sided significance level 0.05

5. Secondary Outcome: Change From Baseline in FSFI Total Score ("Sexual Functioning")
Description: The FSFI total score measures self-reported female sexual functioning covering the major domains arousal, satisfaction, and orgasm, and including lubrication and pain. Possible scores range from 2 to 36, with higher scores indicating better functioning. Change score is calculated by subtracting baseline from later score, with a positive change score indicating increased functioning. This measure is referred to as "sexual functioning" in the protocol.
Time Frame: Baseline (prior to randomization) and 5 and 9 weeks from start of treatment (within 21 days of randomization)
Population: Eligible with baseline data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 78 | 74 | 77
units on a scale
  Week 5: number analyzed (Participants) | 64 | 58 | 61
  Week 5 | 3.84 (7.84) | 4.01 (6.08) | 3.53 (7.48)
  Week 9: number analyzed (Participants) | 61 | 54 | 60
  Week 9 | 3.29 (7.66) | 3.55 (6.63) | 4.70 (8.36)
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Week 5; Test type: Superiority; p = 0.41, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; Week 5; Test type: Superiority; p = 0.35, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 3: Comparison: Bupropion 150 mg vs Placebo; Week 9; Test type: Superiority; p = 0.83, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 4: Comparison: Bupropion 300 mg vs Placebo; Week 9; Test type: Superiority; p = 0.79, t-test, 1 sided — One-sided significance level 0.05

6. Secondary Outcome: Change From Baseline in the Patient Health Questionnaire (PHQ)-4 Score ("Depressive Mood")
Description: The PHQ-4 is a brief screening questionnaire for depression. Possible scores range from 0 to 12, with higher scores indicating more severe depression. Change score is calculated by subtracting baseline from later score, with a negative change score indicating decreased severity of depression. This measure is referred to as "depressive mood" in the protocol.
Time Frame: Baseline (prior to randomization) and 5 and 9 weeks from start of treatment (within 21 days of randomization)
Population: Eligible with baseline data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 79 | 74 | 77
units on a scale
  Week 5: number analyzed (Participants) | 66 | 60 | 62
  Week 5 | -0.44 (1.77) | -0.17 (1.91) | -0.16 (2.29)
  Week 9: number analyzed (Participants) | 65 | 61 | 63
  Week 9 | -0.42 (1.68) | -0.43 (1.86) | -0.43 (2.39)
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Week 5; Test type: Superiority; p = 0.78, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; Week 5; Test type: Superiority; p = 0.51, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 3: Comparison: Bupropion 150 mg vs Bupropion 300 mg; Week 9; Test type: Superiority; p = 0.49, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 4: Comparison: Bupropion 300 mg vs Placebo; Week 9; Test type: Superiority; p = 0.50, t-test, 1 sided — One-sided significance level 0.05

7. Secondary Outcome: Global Impression of Change at 9 Weeks ("Perception of Change")
Description: Participants are asked, "Since beginning the study agent, my desire of sexual intimacy is:" with seven possible answers of "very much better," "moderately better," "a little better," "about the same," "a little worse," "moderately worse," and "very much worse." The first three answers have been categorized as "Better' and the last three answers as "Not Better". This measure is referred to as "perception of change" in the protocol.
Time Frame: 9 weeks from start of study treatment (within 21 days of randomization)
Population: Eligible with data
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 66 | 60 | 63
Participants
  Not Better | 43 | 36 | 43
  Better | 23 | 24 | 20
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Test type: Superiority; p = 0.71, Chi-squared; One-sided significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; Test type: Superiority; p = 0.34, Chi-squared; One-sided significance level 0.05

8. Secondary Outcome: Perception of Risk vs. Benefit at 9 Weeks
Description: Participants are asked, "Were the benefits of this treatment greater than any side effects?"
Time Frame: 9 weeks from start of study treatment (within 21 days of randomization)
Population: Eligible with data
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 67 | 58 | 61
Participants
  No | 37 | 32 | 40
  Yes | 30 | 26 | 21
Statistical Analysis 1: Comparison: Bupropion 150 mg vs Placebo; Test type: Superiority; p = 0.23, t-test, 1 sided — One-sided significance level 0.05
Statistical Analysis 2: Comparison: Bupropion 300 mg vs Placebo; Test type: Superiority; p = 0.25, t-test, 1 sided — One-sided significance level 0.05

9. Secondary Outcome: Number of Participants With a Grade 3 or Higher Adverse Event Over the Course of the Study
Description: Common Terminology Criteria for Adverse Events (version 4) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure.; see Adverse Events Module for specific adverse event data.
Time Frame: Adverse events were evaluated 1,2,5,7, and 9 weeks from start of study treatment (within 21 days of randomization).
Population: Eligible with adverse event data and started study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 77 | 73 | 76
Participants | 4 | 1 | 3

10. Secondary Outcome: Number of Participants With Most Severe Response for Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) at 9 Weeks
Description: Questions refer to the participants' experiences for the past 7 days of a given symptom in terms of frequency (never, rarely, occasionally, frequently, almost constantly), severity (none, mild, moderate, severe, very severe), interference with usual or daily activities (not at all, a little bit, somewhat, quite a bit, very much).
Time Frame: 9 weeks from start of study treatment (within 21 days of randomization).
Population: Eligible with 9 week data
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
Number analyzed (Participants) | 57 | 52 | 56
Participants
  Severity of dry mouth at its worst = very severe: number analyzed (Participants) | 56 | 52 | 56
  Severity of dry mouth at its worst = very severe | 0 | 0 | 0
  Severity of decreased appetite at its worst= very severe | 0 | 0 | 0
  Interference of decreased appetite with usual or daily activities = very much: number analyzed (Participants) | 56 | 51 | 56
  Interference of decreased appetite with usual or daily activities = very much | 0 | 0 | 0
  Frequency of nausea = almost constantly: number analyzed (Participants) | 57 | 51 | 54
  Frequency of nausea = almost constantly | 1 | 0 | 0
  Severity of nausea at its worst = very severe: number analyzed (Participants) | 56 | 50 | 56
  Severity of nausea at its worst = very severe | 0 | 0 | 0
  Severity of constipation at its worst = very severe | 0 | 0 | 0
  Severity of dizziness at its worst = very severe: number analyzed (Participants) | 57 | 52 | 54
  Severity of dizziness at its worst = very severe | 0 | 0 | 0
  Interference of dizziness with usual or daily activities = very much: number analyzed (Participants) | 55 | 51 | 55
  Interference of dizziness with usual or daily activities = very much | 0 | 0 | 0
  Frequency of headache = almost constantly | 0 | 0 | 0
  Severity of headache at its worst = very severe: number analyzed (Participants) | 56 | 51 | 56
  Severity of headache at its worst = very severe | 0 | 1 | 0
  Interference of headache with usual or daily activities = very much: number analyzed (Participants) | 56 | 51 | 56
  Interference of headache with usual or daily activities = very much | 0 | 1 | 0
  Severity of insomnia at it's worst = very severe | 0 | 0 | 1
  Interference of insomnia with usual or daily activities = very much: number analyzed (Participants) | 57 | 51 | 56
  Interference of insomnia with usual or daily activities = very much | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1,2,5,7, and 9 weeks from start of study treatment (within 21 days of randomization).]
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants with adverse event data who started protocol treatment.
Arm/Group | Bupropion 150 mg | Bupropion 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/74 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/77 | 0/73 | 0/76
Other Adverse Events (participants affected / at risk) | 53/77 | 55/73 | 57/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion 150 mg (N=77) | Bupropion 300 mg (N=73) | Placebo (N=76)
Insomnia (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion 150 mg (N=77) | Bupropion 300 mg (N=73) | Placebo (N=76)
Tinnitus (Ear and labyrinth disorders) | 4 | 0 | 2
Constipation (Gastrointestinal disorders) | 23 | 24 | 20
Diarrhea (Gastrointestinal disorders) | 4 | 3 | 8
Dry mouth (Gastrointestinal disorders) | 21 | 30 | 25
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 12 | 14 | 22
Fatigue (General disorders) | 5 | 6 | 5
Pain (General disorders) | 4 | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 13 | 15 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 7
Dizziness (Nervous system disorders) | 9 | 13 | 14
Headache (Nervous system disorders) | 23 | 36 | 30
Tremor (Nervous system disorders) | 4 | 4 | 6
Anxiety (Psychiatric disorders) | 4 | 5 | 3
Depression (Psychiatric disorders) | 4 | 3 | 4
Insomnia (Psychiatric disorders) | 24 | 27 | 29
Libido decreased (Psychiatric disorders) | 1 | 0 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 14
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 4
Hot flashes (Vascular disorders) | 5 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT03180294/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT03180294/ICF_001.pdf